CLINICAL TRIAL: NCT03040232
Title: Clinical Outcomes Following Patellar Dislocation in Young Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2011-1984
Record Dates: First submitted 2017-01-10; First posted 2017-02-02 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Patella Dislocation Recurrent; Patellar Dislocation
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPFl Reconstruction (Experimental): subjects that have had MPFL reconstruction surgery
  Interventions: Other: biomechanical assessment
- Active Controls (Active Comparator): subjects that have not had MPFL reconstruction surgery
  Interventions: Other: biomechanical assessment

INTERVENTIONS:
Other: biomechanical assessment — biomechanical and strength assessment of both groups

SUMMARY:
The purpose of this study is to identify predictors of future injury and disability following LPD. The investigators' long term goal is to improve longitudinal outcomes of athletes with LPD following surgical and non-surgical management. Currently, there is limited information available to clinicians regarding appropriate criteria for returning athletes to sports participation following LPD. The evidence produced by this study will provide necessary information to develop appropriate rehabilitation strategies that may reduce the risk for future patellar instability and associated patellofemoral joint dysfunction and pain.

DETAILED DESCRIPTION:
The basis of the proposed study is to determine the clinical outcomes following lateral patellar dislocation (LPD). Despite surgical and non-surgical interventions, young athletes are at high risk for sustaining subsequent dislocations that magnify the effects of disability. It is suspected that if athletes return to high-level activities and expose their knees to substantial forces without normalized movement strategies, then this may increase the risk for future joint injury. Currently, there are no evidence-based criteria to determine an athlete's readiness for sports activity following LPD. The purpose of this study is to characterize clinical outcomes, function, and neuromuscular control strategies employed by athletes following LPD at the time when they are returning to sports participation.

A prospective, longitudinal study design will be utilized. A cohort of up to 100 athletes (ages 12 - 25 years) who have sustained LPD during sports activities that require jumping, cutting, or pivoting maneuvers will be consecutively recruited from the offices of local orthopaedic surgeons, primary care physicians, and sports physical therapists for this study. Investigators will target a subset of surgically managed athletes and a subset of non-surgically managed athletes with LPD. A cohort of up to 100 individuals without history of knee injury will be recruited from local schools and universities to serve as control participants. Data will be collected to evaluate clinical outcomes, thigh and hip strength, lower body function, balance and neuromuscular control strategies. Clinical outcomes will be assessed using self-report questionnaires and performance-based measures, including hop and agility tests. Thigh and hip strength will be assessed utilizing an isokinetic dynamometer. Lower body function will be assessed using a series of single-leg and double-leg hopping tests. Balance will be assessed utilizing a clinical lower extremity reach test. Neuromuscular control will be evaluated by 3-D motion analysis during running, jumping, and cutting activities. Overall, this study will provide a comprehensive evaluation of athletes following LPD. It will provide important information for the future development of rehabilitation approaches that may maximize clinical outcomes for the at risk population.

ELIGIBILITY:
Inclusion Criteria:

* Participants with LPD who have been managed with non-surgical rehabilitation, pre-surgical rehabilitation, and medial patellofemoral ligament reconstruction (MPFL-R) may be included.
* Participants may be included in this study is they have completed supervised rehabilitation and have been cleared to return to sports participation by their physician.

Exclusion Criteria:

1. lower extremity orthopedic surgeries other than procedures for patellar instability
2. lower extremity injuries within the last 3 months other than patellar dislocation
3. neurological disorders
4. medical conditions that might affect neuromuscular performance.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
change in biomechanical assessment using motion analysis | 6 months
  measure changes in biomechanics between groups using motion analysis with particular interest in knee valgus measures

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Cincinanti Childrens Hospital
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No